CLINICAL TRIAL: NCT05484895
Title: Mobile Health Intervention to Increase HIV Self Testing and Linkage to Services for High-Risk Men in China
Brief Title: Mobile Health Intervention to Increase HIV Testing and Linkage to Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Anhui Medical University (Other); Rutgers University (Other); University of Arkansas (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Don Operario, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00005966; R01MH123352 (NIH)
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: HIV
Keywords: HIV self-testing; Mobile Health; Men who have sex with men; Linkage to care; China
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Intervention Model Description: Intervention involves demonstration of HIV self-testing and access to a mobile health application to promote HIV self-testing, HIV behavioral risk reduction, and linkage to care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WeTest-WeLink intervention (Experimental): Participants will have access to "WeTest-WeLink" application on the WeChat platform, which provides multi-media contents on HIV-related health information, online self-assessments, linkage to providers, data reports, and personal stories, in addition to two-way communication with non-governmental organizations (NGOs), and free, additional HST.
  Interventions: Behavioral: WeTest-WeLink
- Control (Active Comparator): Participants will receive contact information to local NGO to request basic information or receive emergency referrals; have access to "standard" WeChat group; and have free, additional HST.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: WeTest-WeLink — "WeTest-WeLink" application on the WeChat platform provides videos on HIV self-testing and linkage to care; informational articles on HIV, sexually transmitted infections (STI), testing, antiviral treatment (ART), and care; online behavioral self-assessments; linkage to providers; local data reports; stories about coping, wellness, and social support; two-way communication with NGO; and free, additional HST.
  Arms: WeTest-WeLink intervention
Behavioral: Control condition — Contact information of local NGO for emergency referrals; free additional HST.
  Arms: Control

SUMMARY:
This 5-year project will test an mobile health approach to improve HIV self-testing (HST) and linkage to HIV-related care among high-risk men in China. HIV-negative men who have sex with men (MSM) will be randomly assigned to an intervention group: access to WeTest-WeLink (a mobile application-based HIV testing health promotion and risk reduction program), or a control group. Participant HST and sexual risk behaviors will be evaluated at baseline and at 6, 12, and 18 months post-baseline.

DETAILED DESCRIPTION:
The overarching goal of this 5-year research project is to advance the science of mobile health approaches to increase uptake of repeat HIV self-testing (HST) and linkage to HIV-related care with populations that underperform on these steps of the HIV care continuum. The proposed intervention is entitled "WeTest-WeLink" that builds on years of formative work with men who have sex with men (MSM) in China conducted by this team of investigators (R34MH106349), demonstrating promising effects from a pilot RCT and strong indication of intervention acceptability, feasibility, and cultural sensitivity. The intervention uses the "WeChat" mobile app platform, which offers multiple features built into the app that facilitate health information delivery and communication channels (e.g., capacity for private texts, group chats, video sharing, Global Positioning System (GPS), instant messaging, real-time audio and visual communication). Guided by the Information-Motivation-Behavioral (IMB) model and Minority Stress Theory, the study team will employ a user-centered design process to refine and expand app features to support repeat HST uptake, behavioral risk reduction, stigma coping strategies, and self-efficacy to link to HIV care. The study team will use an Effectiveness-Implementation Hybrid Type 1 design consisting of a three site, 2-arm randomized clinical trial (RCT) to test HST and linkage to HIV related care outcomes as well as qualitative research to examine implementation and scalability. The study team will recruit 1,800 HIV negative MSM. Participants will be allocated to the intervention (access to the WeTest-WeLink app) or control group (education about HST and passive referral to HIV care for individuals who test HIV positive). The study team will assess participants at 6, 12, and 18 months to measure intervention effects on primary outcomes of repeated use of HST (including photographic confirmation) and linkage to care for individuals who test HIV-positive. Secondary outcomes include sexual risk behaviors and use of HIV prevention services, and investigators will conduct mediation analysis to examine theoretical mechanisms of behavior change. The study team will qualitatively assess intervention-related process characteristics that enable and/or impede implementation and scalability informed by the Consolidated Framework for Implementation Research (CFIR). This project will provide the first known evidence for a mobile health approach to optimize both HIV testing and linkage to care as part of a single intervention continuum with MSM. Such findings can be crucial for optimizing the care cascade in populations that underutilize HIV services, such as MSM in China and elsewhere in the world where HIV testing and linkage to care services are sub-optimal.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Chinese
* Cis-gender male
* Condomless anal sex with another man in the past 6 months
* Resident in the study location for at least 6 months and no desire to relocate during the study period
* In possession of a mobile "smart" phone with capability to download and use WeChat
* HIV-negative (verified through HIV self-test at enrollment)
* Able to give informed consent

Exclusion Criteria:

* HIV positive at enrollment
* Self-report coercion to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender male
Enrollment: 1800 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Operario, PhD, Principal Investigator — Emory University; Cui Yang, PhD, Principal Investigator — Rutgers University
Locations (3):
- China (3):
  - Wuhan Centers for Disease Control and Prevention, Wuhan, Hubei
  - Suzhou Centers for Disease Control and Prevention, Suzhou, Jiangsu
  - Chengdu Tongle Health Counselling Service Center, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets and a comprehensive data dictionary will be made available for sharing with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available for sharing after data analysis for this study is complete.
Access Criteria: Data will be made available for sharing with researchers, community-based organizations, and advisory committees for the purposes of secondary descriptive or exploratory analysis. Researchers interested in using this data can contact the study PI, Dr. Operario, at don.operario@emory.edu with a brief explanation of the planned analysis.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WeTest-WeLink intervention | Control
Started | 900 | 900
Completed | 837 | 836
Not Completed | 63 | 64
Not completed — Lost to Follow-up | 63 | 64

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WeTest-WeLink intervention | Control | Total
Number analyzed (Participants) | 900 | 900 | 1800
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  18-24 years | 224 | 228 | 452
  25-39 years | 509 | 511 | 1020
  >=40 years | 147 | 161 | 308
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 900 | 900 | 1800
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 900 | 900 | 1800
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 900 | 900 | 1800
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 900 | 900 | 1800

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing HIV Self-Testing
Description: HIV self-testing is assessed by electronic confirmation of HIV self-test result submitted via a mobile app.
Time Frame: Months 6, 12, and 18
Measure: Count of Participants; unit: Participants
Arm/Group | WeTest-WeLink intervention | Control
Number analyzed (Participants) | 900 | 900
Participants
  Month 6 | 878 | 889
  Month 12 | 857 | 875
  Month 18 | 837 | 836

2. Secondary Outcome: Number of Participants With HIV Laboratory Test Results
Description: Linkage to HIV care among study participants who test positive for HIV is measured as confirmation of laboratory test results of cluster of differentiation 4 (CD4) and HIV viral load.
Time Frame: Months 6, 12, and 18
Measure: Count of Participants; unit: Participants
Arm/Group | WeTest-WeLink intervention | Control
Number analyzed (Participants) | 900 | 900
Participants
  Month 6 | 3 | 6
  Month 12 | 6 | 5
  Month 18 | 3 | 5

3. Secondary Outcome: Number of Participants Attending Initial HIV Care Appointment
Description: Linkage to HIV care among study participants who test positive for HIV is measured as confirmation of attendance at an initial HIV care appointment with a local provider.
Time Frame: Months 6, 12, and 18
Measure: Count of Participants; unit: Participants
Arm/Group | WeTest-WeLink intervention | Control
Number analyzed (Participants) | 900 | 900
Participants
  Month 6 | 3 | 6
  Month 12 | 6 | 5
  Month 18 | 3 | 5

4. Secondary Outcome: Number of Participants Receiving Receipt of HIV Confirmatory Test
Description: Linkage to HIV care among study participants who test positive for HIV is measured as confirmation of receipt of an HIV confirmatory test.
Time Frame: Months 6, 12, and 18
Measure: Count of Participants; unit: Participants
Arm/Group | WeTest-WeLink intervention | Control
Number analyzed (Participants) | 900 | 900
Participants
  Month 6 | 3 | 6
  Month 12 | 6 | 5
  Month 18 | 3 | 5

5. Other Pre Specified Outcome: Number of Participants Using HIV Prevention Services
Description: Participants are asked to report whether or not they have used any HIV prevention services.
Time Frame: Months 6, 12, and 18
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Number of Participants Reporting Substance Use
Description: HIV risk behavior is assessed by participants self-reporting alcohol or drug use prior to or during sexual episodes during the past 3 months.
Time Frame: Months 6, 12, and 18
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Number of Participants Reporting Condomless Anal Sex
Description: HIV sexual risk is assessed as participants' self-report of condomless anal sex.
Time Frame: Months 6, 12, and 18
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the duration of the study, up to 18 months post-intervention.
Arm/Group | WeTest-WeLink intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/900 | 0/900
Serious Adverse Events (participants affected / at risk) | 0/900 | 0/900
Other Adverse Events (participants affected / at risk) | 0/900 | 0/900

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT05484895/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT05484895/ICF_000.pdf